CLINICAL TRIAL: NCT07334197
Title: Effect of Melatonin in Peripartum Cardiomyopathy
Brief Title: Effect of Melatonin on Left Ventricular Reverse Remodeling and Inflammation in Peripartum Cardiomyopathy
Acronym: MEL-PPCM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Reem Alaa Abdel Samie, Teacher assistant in faculty of pharmacy, delta university for science and technology, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEL-PPCM
Record Dates: First submitted 2026-01-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Ppm, Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies | interventions — Melatonin; Selenium

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of four groups to evaluate effects on left ventricular remodeling and inflammation:
  Standard heart failure therapy alone (Control) Standard therapy + Melatonin Standard therapy + Selenium Standard therapy + Melatonin + Selenium
Who Masked: Participant, Care Provider
Masking Description: participants, care providers are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control (Active Comparator): Participants receive standard guideline-directed heart failure therapy alone. Therapy includes beta-blockers, ACE inhibitors/ARBs/ARNI, diuretics, and mineralocorticoid receptor antagonists as clinically indicated for 3 months.
  Interventions: Drug: Placebo
- Melatonin (Experimental): Participants receive standard heart failure therapy plus melatonin 10 mg orally once daily at bedtime for 3 months.
  Interventions: Drug: Melatonin 10 MG
- Selenium (Experimental): Participants receive standard heart failure therapy plus selenium 100 μg orally once daily for 3 months.
  Interventions: Drug: Selenium
- Melatonin + Selenium (Experimental): Participants receive standard heart failure therapy plus melatonin 10 mg orally once daily at bedtime and selenium 100 μg orally once daily for 3 months.
  Interventions: Drug: Melatonin 10 MG; Drug: Selenium

INTERVENTIONS:
Drug: Melatonin 10 MG — Melatonin 10 mg orally once daily at bedtime for 3 months, administered in addition to standard guideline-directed heart failure therapy. Melatonin is a naturally occurring hormone with antioxidant and anti-inflammatory effects, aimed at improving left ventricular reverse remodeling and reducing systemic inflammation in patients with peripartum cardiomyopathy.
  Other Names: melatonin
  Arms: Melatonin; Melatonin + Selenium
Drug: Selenium — Selenium 100 μg orally once daily for 3 months, administered in addition to standard guideline-directed heart failure therapy. Selenium is an essential trace element with antioxidant properties, hypothesized to reduce inflammation and improve cardiac recovery in peripartum cardiomyopathy.
  Arms: Melatonin + Selenium; Selenium
Drug: Placebo — control group takes Placebo
  Arms: control

SUMMARY:
This randomized, controlled clinical trial investigates the potential cardioprotective effects of melatonin in women diagnosed with peripartum cardiomyopathy (PPCM). The study aims to determine whether melatonin supplementation improves left ventricular (LV) function, promotes reverse remodeling, and reduces systemic inflammation. Participants receive standardized heart failure therapy with or without adjunctive melatonin, and outcomes are assessed using echocardiographic parameters (including LVEF, LV dimensions, and global longitudinal strain) and inflammatory biomarkers (e.g., CRP, IL-6, TNF-α). The study hypothesizes that melatonin's antioxidant and anti-inflammatory properties will enhance cardiac recovery, improve functional capacity, and potentially reduce morbidity in PPCM patients.

DETAILED DESCRIPTION:
Peripartum cardiomyopathy is a rare but serious cause of heart failure in late pregnancy or early postpartum, often associated with significant morbidity. Current treatment primarily relies on guideline-directed heart failure therapy, but adjunctive interventions to accelerate ventricular recovery and mitigate inflammation remain limited.

Melatonin, a naturally occurring hormone, has antioxidant, anti-inflammatory, and cardioprotective effects demonstrated in preclinical and clinical heart failure studies. This trial evaluates melatonin as a complementary therapy to improve LV remodeling in PPCM.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with peripartum cardiomyopathy Age between 18-45 years. Left ventricular ejection fraction (LVEF) ≤ 45% at baseline. Able to provide written informed consent.

Exclusion Criteria:

* History of pre-existing cardiomyopathy or significant structural heart disease before pregnancy.

Severe renal (eGFR <30 mL/min/1.73m²) or hepatic dysfunction. Active infection or inflammatory disease that may confound biomarker measurements.

Known hypersensitivity to melatonin or selenium. Current participation in another interventional clinical trial. Inability to comply with study protocol or follow-up visits.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female only, as peripartum cardiomyopathy occurs in women during late pregnancy or postpartum.
Enrollment: 25 (Estimated)
Dates: Start 2026-12-20 (Estimated); Primary Completion 2029-12-20 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline and 3 months
  Absolute change in LVEF measured by transthoracic echocardiography from baseline to 3 months. LVEF will assess left ventricular systolic function and reverse remodeling in participants receiving melatonin, selenium, or combination therapy compared to standard therapy alone.
Change in Left Ventricular End-Diastolic Dimension (LVEDD) | Baseline and 3 months
  Absolute change in LVEDD measured by echocardiography from baseline to 3 months to evaluate structural remodeling.
Global Longitudinal Strain (GLS) Improvement | Baseline and 3 months
  Change in GLS (%) assessed by speckle-tracking echocardiography from baseline to 3 months to assess myocardial contractility.

SECONDARY OUTCOMES:
Change in Inflammatory Biomarkers | Baseline and 3 months
  Absolute changes in serum CRP, IL-6, and TNF-α from baseline to 3 months. These markers assess systemic inflammation and potential anti-inflammatory effects of interventions.
Functional Capacity | Baseline and 3 months
  Change in distance walked in the 6-minute walk test (6MWT) from baseline to 3 months to evaluate improvement in exercise tolerance.